CLINICAL TRIAL: NCT03284528
Title: Does Placenta Pathology Predict Outcome of Neonates With Hypoxic Ischemic Encephalopathy?"
Status: Completed | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-00912
Record Dates: First submitted 2017-09-13; First posted 2017-09-15 (Actual); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Asphyxia Neonatorum
MeSH Terms: conditions — Asphyxia Neonatorum | interventions — Cryotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: hypothermia therapy — newborn infants with hypoxic-ischaemic encephalopathy are cooled for 72 hours with a target temperature of 33-34°C (whole body cooling).

SUMMARY:
The histology of the placenta of newborn infants with perinatal asphyxia and hypoxic-ischaemic encephalopathy is analysed. There will be an evaluation if placenta could be a biomarker for neurodevelopmental outcome at 18-24 months of age.

ELIGIBILITY:
Inclusion Criteria:all newborn infants with APGAR <5 at 10minutes, pH<7.0, lactate >12mmol/L, base excess >16, resuscitation >10min after birth, gestational age >35 weeks and an encephalopathy -

Exclusion Criteria:

-

Ages: 1 Day to 4 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All newborn infants with a gestational Age >35 weeks, fulfilling the inclusion criteria of perinatal asphyxia and hypoxic-ischaemic encephalopathy, born in Switzerland and treated in the University Hospital of Zurich with hypothermia therapy after birth
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
neurodevelopmental outcome at 18-24 month of Age | 7 years
  The investigators will analyse if there is a correlation of placenta histology and neurodevelopmental outcome

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Brotschi, Principal Investigator — University Childrens's hospital of Zurich
Locations (1):
- University Children's hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No